CLINICAL TRIAL: NCT02964234
Title: Empowering Latinas to Obtain Breast Cancer Screenings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: The Resurrection Project (Other); Juan Diego Centro Comunitario (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Yamile Molina, Assistant Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2015-1246; K01CA193918 (NIH)
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Breastcancer; Breast Diseases
Keywords: Mammography Screening; Latinas; Breast cancer disparities
MeSH Terms: conditions — Breast Diseases | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empowerment (Experimental): Behavior: Empowerment
  Interventions: Behavioral: Empowerment
- Education (Experimental): Behavior: Education
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Empowerment — Three group sessions (breast cancer education; communication; volunteerism) 1.5 hours 3 times across 3 weeks
  Arms: Empowerment
Behavioral: Education — Three group sessions (breast cancer education; diet; physical activity) 1.5 hours 3 times across 3 weeks
  Arms: Education

SUMMARY:
The participatory-based project will quantify the 'added benefit' of an empowerment intervention relative to an education intervention for 150 Latinas on the following outcomes: women's adherence to breast cancer screening guidelines; women's psychosocial facilitators (self-efficacy, norms, support, and knowledge); and women's dissemination of breast health messages throughout their social network. The empowerment intervention will train Latinas in how to discuss breast health with their family and friends and volunteer in local breast health promotion programs. Academic, clinician, and community partners will work together throughout intervention development and evaluation.

DETAILED DESCRIPTION:
Latinas suffer disproportionately from breast cancer relative to non-Latina Whites (NLWs), including late stage detection. While there have been controversies in breast cancer screening, non-adherence to guideline-concordant screening continues to be a major modifiable determinant of breast cancer outcome disparities. Thus, increasing participation in breast cancer screening among Latinas, especially care that corresponds with clinical and academic guidelines, is a public health priority. Participatory approaches are popular methods to improve screening within this group and have included approaches that 1) deliver education to non-adherent Latinas and 2) train community health advocates (community health workers, breast cancer survivors) to engage in breast health promotion. The second approach (empowerment interventions) concerns training participants to engage in social outreach (e.g., having conversations with family and friends about breast health) and volunteering (e.g., helping in health fairs, engaging in civic campaigns about breast cancer programs). Patient activation and volunteerism literature suggest that empowerment interventions may have 'added value' for participants themselves over delivering education in terms of preventive health psychosocial factors and practices. Relative to education interventions, empowerment interventions may also affect women's networks, as they may be more likely to disseminate evidence-based breast health promotion among their family and friends. To date, little research has compared interventions' effects on individual-level outcomes or used formal social network analysis to examine network effects. The proposed work adds to the literature through empirically comparing two approaches (education versus empowerment) on three sets of outcomes: 1) women's own screening, 2) women's own self-efficacy, norms, support, knowledge; and 3) women's networks (measured by egocentric analysis). I will lead this work and will benefit from the collective expertise and resources of my mentors (Drs. Ferrans, Mermelstein, Geller) and collaborators (Dr. Schneider, The Resurrection Project, Metropolitan Chicago Breast Cancer Task Force, Sinai Urban Health Institute, University of Illinois Cancer Center). Aim 1 intervention development will be accomplished through continuous stakeholder engagement and specifically through meetings and focus groups with a bilingual, bicultural community advisory engagement board (CEAB), UICC radiologists and target participants (non-adherent Latinas). We have already begun this process and are obtaining formative data. After we develop intervention materials, a pilot trial will be conducted with an area-level treatment control group design in Chicago. Participants will be 150 Latinas with no history of health volunteerism, residence in one of two targeted areas, and non-adherence to US Preventive Services Task Force screening guidelines. Aim 1 intervention evaluation will involve an analysis to compare differences in receipt of a medical record-confirmed screening within six months of participating in the study. Aim 2 will be an analysis to compare interventions' effects on self-efficacy, norms, support, knowledge across three time points - pre-intervention, immediately post-intervention, and six months post-intervention. Aim 3 will be a social network analysis, specifically egocentric, to compare interventions' effects on breast health, network size, and network density as well as will number of peers referred to the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 52-75 years old;
* Identification as Latina/Hispanic/Chicana female;
* Residence in Pilsen, Little Village, East Side or South Chicago;
* No history of health volunteerism;
* No history of breast cancer; and
* Lack of a mammogram within the last two years

Exclusion Criteria:

* Not meeting all inclusion criteria;
* Women will be excluded if they participated in formative focus groups

Ages: 52 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yamile Molina, PhD, Principal Investigator — University of Illinois at Chicago
Locations (3):
- United States (3):
  - The Resurrection Project, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Juan Diego Centro Comunitario, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
After major study findings have been accepted for publication, Dr. Molina will develop an anonymized data set (i.e., no personally identifiable information) available to qualified scientists upon request. Data will only be made available to scientists who complete a data-sharing agreement that indicates: 1) commitment to using the data only for research purposes and not to identify any individual participant; 2) commitment to securing data using appropriate computer technology; and 3) commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol
Time Frame: Data will become available 6 months after publication of the primary outcome papers.
Access Criteria: The study protocol will be shared upon reasonable request by interested researchers. IRB approval will be required before data are released.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Empowerment | Education
Started | 76 | 69
Completed | 54 | 56
Not Completed | 22 | 13
Not completed — Lost to Follow-up | 22 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Empowerment | Education | Total
Number analyzed (Participants) | 76 | 69 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.05 (6.29) | 61.28 (6.36) | 61.16 (6.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 69 | 145
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 69 | 145
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 69 | 145
Insurance [Count of Participants; unit: Participants] | 24 | 40 | 64
Mammogram 4+ years ago [Count of Participants; unit: Participants] | 22 | 30 | 52
Mammography intention within next year [Count of Participants; unit: Participants] | 48 | 40 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Have Obtained Breast Cancer Screening
Description: Receipt of mammogram based on medical records and self report within 6 months of baseline survey (Yes or No)
Time Frame: 6 months
Population: Complete case analysis used - only participants who were retained until 6 month follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Empowerment | Education
Number analyzed (Participants) | 54 | 56
Participants | 49 | 29
Statistical Analysis 1: Comparison: Empowerment vs Education; We conducted logistic regressions, clustering by cohort, given both interventions used a group format, and adjusting for age, education, income, insurance status, baseline mammography history, and baseline mammography intention. The null hypothesis was there would be no study arm differences. A priori power analysis suggested that a sample size of 150, assuming alpha = .05, power = .80 would lead us to detect medium/large effects (OR = 2.8); Test type: Superiority; p = .005, Regression, Logistic — We clustered by cohort, given both interventions used a group format, and adjusted for age, socioeconomic status (education, income, insurance status) baseline mammography history, and baseline mammography intention; Odds Ratio (OR) = 10.59, 95% CI 2-sided [2.01 to 56.31]

2. Other Pre Specified Outcome: Changes in Psychosocial Facilitators of Screening Survey Measures
Description: Total scores/ranges are used. No subscales used. Knowledge - 5 items (Williams et al., 2011). Range for the change scores (baseline to 6-months) is -5 to 5. Higher scores represent a better outcome.
  Cultural beliefs - Ferrans cultural beliefs scale (Ferrans et al., 2007). Range for the change scores (baseline to 6-months) is -17 to 17. Higher scores represent a worse outcome.
  Breast cancer-specific self-efficacy - Mammography-Specific Self-Efficacy Scale (Champion, Skinner, & Menon, 2005). Range for the change scores (baseline to 6-months) is -26 to 26. Higher scores represent a better outcome.
  Positive breast cancer screening norms - 6 items ( Molina et al., 2015). Range for the change scores (baseline to 6-months) is -12 to 12. Higher scores represent a better outcome.
  Breast cancer supportive social network size questions comprised an 8-item version of Berkman-Syme index. Range for the change scores (baseline to 6-months) is -25 to 25. Higher scores represent a better outcome.
Time Frame: Baseline and 6 months
Population: This is a complete case analysis for outcome data, with all available data being used for participants who completed the 6-month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Empowerment | Education
Number analyzed (Participants) | 54 | 56
units on a scale
  Knowledge | 0.98 (1.60) | 1.37 (1.69)
  Cultural Beliefs | -1.36 (2.94) | -2.41 (3.13)
  Self-Efficacy | 1.02 (4.67) | -1.00 (5.99)
  Social Norms | 0.25 (2.42) | 0.32 (2.94)
  Supportive Network size | 1.38 (4.66) | 5.85 (2.11)
Statistical Analysis 1: Comparison: Empowerment vs Education; Analyses were conducted using GEE with an exchangeable correlation structure and a gamma distribution with log link. All models included study arm, time, and the study arm*time. Covariates included age, education, and mammography history. With 150 Latinas, alpha = 0.05, power = 0.80, ICC = 0.0-0.05, we expected to detect small/medium interaction effects; Test type: Superiority; p = 0.03, Regression, Linear; With GEE. Models had exchangeable correlation structure, a gamma distribution, and log link; Slope = -0.19, 95% CI 2-sided [-0.34 to -0.04]

3. Other Pre Specified Outcome: Number of Individuals to Whom Participants Exchanged Information About Breast Cancer Screening.
Description: This was an open-ended questionnaire, based on the Burt Social Network Instrument. Higher numbers represent better outcomes.
Time Frame: 6 months
Population: Complete case analysis used, wherein we focus on participants who completed the 6-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: family/friends engaged
Arm/Group | Empowerment | Education
Number analyzed (Participants) | 54 | 56
family/friends engaged | 8.27 (6.17) | 5.81 (12.58)
Statistical Analysis 1: Comparison: Empowerment vs Education; We used ordinal regression, given the non-normal distribution revealed by preliminary analyses. Analyses clustered by cohort and adjusted for age, SES (education, income, insurance), mammography history, mammography intention, and baseline supportive breast cancer social network size. Power analyses suggested that with 150 Latinas, alpha = .05, power = .80, we would be able to detect a small effect (Cohen's f = 0.05); Test type: Superiority; p < 0.0001, Ordinal regression — Analyses clustered by cohort and adjusted for age, SES (education, income, insurance), mammography history, mammography intention, and baseline supportive breast cancer social network size; Odds Ratio (OR) = 6.15, 95% CI 2-sided [2.82 to 13.32]

ADVERSE EVENTS:
Time Frame: Data were collected for up to 6 months per participant.
Description: We used standard definitions of adverse and serious adverse events.
Arm/Group | Empowerment | Education
All-Cause Mortality (participants affected / at risk) | 0/76 | 3/69
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/69
Other Adverse Events (participants affected / at risk) | 0/76 | 0/69

LIMITATIONS AND CAVEATS:
There are several limitations to this study, including a small sample, use of non-probability based sampling strategies, and non-randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT02964234/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT02964234/ICF_001.pdf